CLINICAL TRIAL: NCT01213628
Title: Intraoperative Local Insufflation of Humidified Warmed CO2 Increases Core and Open Wound Temperatures? - A Randomized Clinical Trial
Brief Title: Local CO2 Increases Core and Wound Temperature
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Jan van der Linden, Professor, Karolinska Institute / Karolinska University Hospital, Stockholm, Sweden
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: Buk1
Record Dates: First submitted 2010-10-01; First posted 2010-10-04 (Estimated); Last update posted 2010-10-04 (Estimated); Status verified 2010-10

CONDITIONS: Hypothermia
Keywords: abdominal surgery; hypothermia; wound desiccation; warming
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Standard heating (Experimental): Standard intraoperative warming measures including heated sheets, heating with forced warmed air, warming of fluids, and insulation of limbs and head.
  Interventions: Device: humidified warmed CO2

INTERVENTIONS:
Device: humidified warmed CO2 — Additional insufflation of humidified carbon dioxide (approx. 30ºC, approx. 80-100% relative humidity) via a simple humidifier (sterile water in plastic bottle) connected to a gas diffuser (Cardia Innovation AB) that is able to create a local atmosphere of 100% carbon dioxide (humidified) in the wound cavity.
  Other Names: CO2; Carbondioxide

SUMMARY:
Eighty adult patients undergoing open colon surgery will be randomized to either:standard warming measures or to additional insufflation of humidified carbon dioxide in the open wound cavity during major abdominal surgery.

PRIMARY AIM is to test if core and local temperature can be increased.

DETAILED DESCRIPTION:
Eighty adult patients undergoing open colon surgery will be randomized to either:

standard warming measures including heating sheets, warming of fluids, and insulation of limbs and head, or to additional insufflation of humidified carbon dioxide (approx. 30ºC, approx. 80-100% relative humidity) via a simple humidifier (sterile warmed water) connected to a gas diffuser (Cardia Innovation AB) that is able to create a local atmosphere of 100% carbon dioxide (humidified ) in the open wound cavity.

PRIMARY AIM The primary aim of this study is to evaluate if humidified carbon dioxide insufflated into an open surgical wound can be used to warm the core, open wound cavity, and the wound edges during major abdominal surgery.

SECONDARY AIMS Secondary aims are to evaluate possible differences between the groups regarding complications and clinical differences including histological signs.

ELIGIBILITY:
Inclusion Criteria:

* major open abdominal surgery (colon surgery) in adults patient signed informed consent

Exclusion Criteria:

* acute surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2007-03; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Temperature | up to 12 hours after start of surgery
  Core temperature measurement via tympanic thermometer, wound temperatures via an infrared camera

SECONDARY OUTCOMES:
Time to extubation | up to 30 days after surgery
Intraoperative bleeding | up to 12 hours after start of surgery
  ml
Hospital stay | up to 60 days after surgery
  days in hospital

CONTACTS AND LOCATIONS:
Overall Officials: Jan A van der Linden, MD PhD, Principal Investigator — Karolinska Institute, Karolinska University Hospital
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

REFERENCES:
- [Background] Persson M, van der Linden J. Perioperative cooling to prevent adhesion formation may be counterproductive for the clinical outcome. Hum Reprod. 2009 Nov;24(11):2965; author reply 2966-7. doi: 10.1093/humrep/dep326. Epub 2009 Sep 9. No abstract available. PMID 19740898
- [Background] Persson M, van der Linden J. Intraoperative field flooding with warm humidified CO2 may help to prevent adhesion formation after open surgery. Med Hypotheses. 2009 Oct;73(4):521-3. doi: 10.1016/j.mehy.2009.06.009. Epub 2009 Jul 8. PMID 19589645
- [Background] Persson M, van der Linden J. Intraoperative CO2 insufflation can decrease the risk of surgical site infection. Med Hypotheses. 2008;71(1):8-13. doi: 10.1016/j.mehy.2007.12.016. Epub 2008 Mar 4. PMID 18304752
- [Background] Persson M, van der Linden J. Can wound desiccation be averted during cardiac surgery? An experimental study. Anesth Analg. 2005 Feb;100(2):315-320. doi: 10.1213/01.ANE.0000140243.97570.DE. PMID 15673849
- [Background] Persson M, Svenarud P, Flock JI, van der Linden J. Carbon dioxide inhibits the growth rate of Staphylococcus aureus at body temperature. Surg Endosc. 2005 Jan;19(1):91-4. doi: 10.1007/s00464-003-9334-z. Epub 2004 Nov 11. PMID 15529188
- [Background] Persson M, Elmqvist H, van der Linden J. Topical humidified carbon dioxide to keep the open surgical wound warm: the greenhouse effect revisited. Anesthesiology. 2004 Oct;101(4):945-9. doi: 10.1097/00000542-200410000-00020. PMID 15448528
- [Background] Persson M, Svenarud P, van der Linden J. What is the optimal device for carbon dioxide deairing of the cardiothoracic wound and how should it be positioned? J Cardiothorac Vasc Anesth. 2004 Apr;18(2):180-4. doi: 10.1053/j.jvca.2004.01.024. PMID 15073708
- [Background] Sessler DI. New surgical thermal management guidelines. Lancet. 2009 Sep 26;374(9695):1049-50. doi: 10.1016/S0140-6736(09)61686-X. No abstract available. PMID 19782858
- [Background] Sessler DI. Temperature monitoring and perioperative thermoregulation. Anesthesiology. 2008 Aug;109(2):318-38. doi: 10.1097/ALN.0b013e31817f6d76. PMID 18648241
- [Derived] Frey JM, Janson M, Svanfeldt M, Svenarud PK, van der Linden JA. Intraoperative local insufflation of warmed humidified CO(2) increases open wound and core temperatures: a randomized clinical trial. World J Surg. 2012 Nov;36(11):2567-75. doi: 10.1007/s00268-012-1735-5. PMID 22868970